CLINICAL TRIAL: NCT05534282
Title: Interaction-focused Music Therapy With Cancer Affected Children and Their Significant Others: a Randomized Controlled Feasibility Study With Subsequent Intervention (INMUT)
Brief Title: Music Therapy With Cancer Affected Children and Their Families
Acronym: INMUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Heidehof Foundation Stuttgart (Unknown); Community Hospital Herdecke (Unknown); Nordoff/Robbins Music Therapy Center Witten (Unknown); Interprofessional Graduate Programm in Integrative Medicine IGIM (Unknown)
Responsible Party: Principal Investigator, Constance Boyde, cand. Dr., University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INMUT
Record Dates: First submitted 2022-08-08; First posted 2022-09-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Cancer
Keywords: pediatrics oncology; music therapy; children; family; significant others
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interaction-focused Music Therapy with Children and Significant Others (INMUT-KB) (exp. group) (Experimental): Interaction-focused music therapy with children with cancer and their significant others, delivered by trained music therapists
  Interventions: Behavioral: Interaction-focused Music Therapy with Children and Significant Others (INMUT-KB) (exp. group)
- Music Therapy with Children (MUT-K) (exp. group) (Experimental): Interaction-focused music therapy with children with cancer without the involvement of significant others, delivered by trained music therapists.
  Interventions: Behavioral: Music Therapy with Children (MUT-K) (exp. group)
- Interaction-focused Music Therapy with Children and Significant Others (WG-KB) (control group) (Experimental): Study participants randomized to this group receive the intervention INMUT 10 weeks after the experimental groups.
  Interventions: Behavioral: Interaction-focused Music Therapy with Children and Significant Others (WG-KB) (control group)

INTERVENTIONS:
Behavioral: Interaction-focused Music Therapy with Children and Significant Others (INMUT-KB) (exp. group) — Interaction-focused music therapy with children with cancer and their significant others, delivered by trained music therapists.
  Arms: Interaction-focused Music Therapy with Children and Significant Others (INMUT-KB) (exp. group)
Behavioral: Music Therapy with Children (MUT-K) (exp. group) — Interaction-focused music therapy with children with cancer without the involvement of significant others, delivered by trained music therapists.
  Arms: Music Therapy with Children (MUT-K) (exp. group)
Behavioral: Interaction-focused Music Therapy with Children and Significant Others (WG-KB) (control group) — Study participants randomized to this group receive the intervention INMUT 10 weeks after the experimental groups.
  Arms: Interaction-focused Music Therapy with Children and Significant Others (WG-KB) (control group)

SUMMARY:
Background: Pediatric oncology patients and their families are in an existentially threatening situation for which music therapy has proven as a cross-linguistic field of action: the creative act of making music offers the possibility of strengthening individual competences and makes socio-psycho-biological conflicts tangible in a very direct way. Although music therapy is an established component of multimodal care and the inclusion of significant others in the therapy setting is recommended, there has been little clinical research on music therapy interaction processes in the family system. The researchers have designed a randomized controlled pilot trial (INMUT) that specifically addresses family interaction in a multi-person setting.

Methods: The examiners investigate the efficacy of music therapy interventions involving the parent-child dyad (INMUT-KB, n=16) compared to music therapy interventions involving only the child (MUT-K, n=16) and a waiting group without intervention (WG, n=10).

Research questions: 1) Does the parent-child interaction improves in mutual attunement, nonverbal communication, and emotional parental response? 2) Are there effects on quality of life, psychosocial and psychosomatic impairments, and system-related level of functioning? Evaluation tools: Primary goals will be assessed by the music therapy-based Assessment of parent-child interaction (APCI) pre and post. The secondary objectives will be assessed by self-reports in form of the psychometric questionnaires KINDL, Experience in Social Systems Questionnaire (EXIS), Burden Assessment Scale (BAS) and Symptom Checklist-K-9 (SCL-9K) pre, post and follow up.

Discussion: The investigators hope for an improvement of the primary and secondary endpoints through participation in music therapy as a basis for a needs-oriented accompaniment of families.

ELIGIBILITY:
Inclusion Criteria, Children:

* cancer diagnosis
* inpatient (e.g. GKH)
* no cognitive and auditory dysfunction

Exclusion Criteria, Children:

* Serious comorbidity with impairment of brain-organic functions
* BMI<14
* serious physical comorbidity that does not allow specific assessment of psychosomatic constructs with certainty
* withdrawal of informed consent

Inclusion Criteria, Important Reference Persons:

- e.g. father, mother, siblings

Exclusion Criteria, Important Reference Persons:

- withdrawal of consent

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Parent-Child Interaction (APCI) | Baseline, Change in 10th hour of intervention
  The APCI captures child-reference interaction using mutual attunement, nonverbal communication, and emotional parental response. The diagnostic music therapy intervention sessions are conducted and evaluated by external, blinded, APCI-certified raters.

SECONDARY OUTCOMES:
KINDL-Children/YouthVersion, Modul Oncology | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  The KINDL uses 40 items to assess the psychological well-being, social relationships, physical functioning, and daily activities during the daily activities within the last week.
Symptom Checklist-K-9 (SCL-9k) | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  The "Short Form Symptom Checklist" (SCL-9k) captures impairment using 9 statements about somatization, obsessiveness, social insecurity, depressiveness, anxiety, aggressiveness, phobic anxiety, paranoia, and psychoticism.
Experience in Social Systems Questionnaire (EXIS) | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  EXIS, the "Questionnaire on Experience in Private Social Systems", measures on basis of 12 items the degree of belonging, autonomy, accord, and confidence in the social system described as important within the past 2 weeks.
Burden Assessment Scale (BAS) | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  The BAS uses 19 items to survey personal stress, feelings of guilt, the need to interrupt and postpone important matters, and a changed and altered perspective of time in relation to the symptoms displayed by the ill relatives within the last 6 months.
Wittener Ressources Questionnaire (WIRF) | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  WIRF captures resources on the basis of three domains of coping with general life experiences, difficult situations in the past, and current problems, using 12 items each. We will use the domain of coping with general life esperiences.
Goal Attainement Scale (GAS) | Baseline, Change in 10th hour of intervention, Change in 3 months after intervention
  GAS captures in free text the subjective goals of children and their significant others. These are classified using the Bern Inventory for Therapy (BIT-T): (1) coping with specific problems and symptoms, (2) interpersonal goals, (3) well-being, (4) existential issues, (5) personal growth, (6) residual category.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Längler, Prof. Dr., Principal Investigator — Gemeinschaftskrankenhaus Herdecke; Dominik Schneider, Prof. Dr., Principal Investigator — Klinikum Dortmund; Michael Paulussen, Prof. Dr., Principal Investigator — Vestische Kinderklinik Datteln
Locations (3):
- Germany (3):
  - Vestische Kinderklinik Datteln, Datteln
  - Klinikum Dortmund, Dortmund
  - Gemeinschaftskrankenhaus Herdecke, Herdecke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunger C, Hilzinger R, Klewinghaus L, Deusser L, Sander A, Mander J, Bents H, Ditzen B, Schweitzer J. Comparing Cognitive Behavioral Therapy and Systemic Therapy for Social Anxiety Disorder: Randomized Controlled Pilot Trial (SOPHO-CBT/ST). Fam Process. 2020 Dec;59(4):1389-1406. doi: 10.1111/famp.12492. Epub 2019 Oct 27. PMID 31657011
- [Background] Hunger, C. (2020). Familienaufstellung als Einzelintervention im Gruppensetting bei chronisch-psychosozialen Konflikten: Randomisiert-kontrollierte Wirksamkeitsstudie mit Katamnesen von 2 Wochen bis 5 Jahre. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie, 68(4), 263-273.
- [Background] Hunger C, Bornhauser A, Link L, Geigges J, Voss A, Weinhold J, Schweitzer J. The Experience in Personal Social Systems Questionnaire (EXIS.pers): Development and Psychometric Properties. Fam Process. 2017 Mar;56(1):154-170. doi: 10.1111/famp.12205. Epub 2016 Feb 8. PMID 26858173
- [Background] Boyde C, Linden U, Boehm K, Ostermann T. The Use of Music Therapy During the Treatment of Cancer Patients: A Collection of Evidence. Glob Adv Health Med. 2012 Nov;1(5):24-9. doi: 10.7453/gahmj.2012.1.5.009. Epub 2012 Nov 1. PMID 27257528
- [Background] Ostermann, T., Boyde, C., & Linden, K. (2012). Music therapy in the treatment of cancer patients: A systematic review. BMC Complementary and Alternative Medicine, 12(Suppl1): P327.
- [Derived] Boyde C, Berger B, Langler A, Neugebauer L, Jacobsen SL, Swanick R, Gaebel C, Schneider D, Bernbeck B, Paulussen M, Ostermann T, Hunger-Schoppe C. Interaction-focused music therapy with cancer-affected children and their significant others: a randomized controlled feasibility study with subsequent intervention (INMUT). Pilot Feasibility Stud. 2024 May 28;10(1):86. doi: 10.1186/s40814-024-01490-8. PMID 38807165